CLINICAL TRIAL: NCT07125001
Title: The Influence of Mango-Derived Intestinal Microbial Metabolites on Gut Permeability, Inflammation, and Cardiometabolic Health Markers in Hispanic/Latino Adolescents
Brief Title: Mango Intake and Gut and Cardiometabolic Health in Hispanic/Latino Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1939453
Record Dates: First submitted 2025-07-07; First posted 2025-08-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cardiometabolic Health Indicators; Vascular Function in Healthy Volunteers; Inflammation
Keywords: mango; cardiometabolic; adolescents; microbiome
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango arm (Experimental): Ataulfo Mango intake
  Interventions: Other: Ataulfo mango
- No mango intake (No Intervention): 4 weeks of no mango intake

INTERVENTIONS:
Other: Ataulfo mango — 4 weeks of Ataulfo mango intake
  Arms: Mango arm

SUMMARY:
Mangos contain a number of nutrients that may improve gut and metabolic health. The purpose of this research is to see how eating mangos every day for 4 weeks instead of snacks high in calories and low in nutrients such as cookies, crackers, chips, and candy can impact adolescent health.

DETAILED DESCRIPTION:
This study will record the functional and metabolic effects of daily mango intake, incorporated into the habitual diets of Hispanic/Latino adolescent children. This racial group is considered the most significant minority in the US, accounting for 19.1% of the population. The proposed study design allows for comparing baseline metabolic and physiological function to the real-world situation of adding a new snack food to a child in the major minority group in the US habitual diet. Moreover, the study design will allow the assessment of dietary changes in an understudied population at increased cardiovascular risk due to the high prevalence of overweight and obesity. Collectively, these analyses will help identify the complex relationships of mango-derived nutrients and microbial metabolites to physiologic response.

Twenty-five (12-19 years of age) adolescents will be enrolled in a randomized, controlled 2-arm crossover dietary intervention trial. Participants will be randomized to consume either ¾ cups of mango or continue their habitual diet for 4 weeks, followed by a 4-week washout period before crossing over to the alternate group. The mango flesh will be cut into uniform chunks (2-3 cm) and portioned into individual servings that can be consumed either as-is or blended into a smoothie.

ELIGIBILITY:
Inclusion Criteria:

* - Male or Female 12-19 years old
* BMI ≥ 85th percentile (https://www.bcm.edu/bodycomplab/BMIapp/BMI-calculator-kids.html)
* Self-reported Hispanic/Latino
* Subject is willing and able to comply with the study protocols
* Subject is willing to consume the test products
* Female-specific criteria: if menstruating, eumenorrheic (regular monthly menstrual cycles of 25-30-days in length)
* Access to a smartphone or tablet at least 1x / day and willing to take pictures associated with the products to be consumed in the study

Exclusion Criteria:

* - Reported food allergies.
* Currently taking prescription drugs, with the exception of asthma inhalers, which are allowed
* BMI <85th percentile (https://www.bcm.edu/bodycomplab/BMIapp/BMI-calculator-kids.html)
* Current participation in a moderate or high-intensity daily exercise routine
* Self-reported disease, serious illness, or who are currently under acute medical care.
* Currently taking prescription drugs.
* Any supplement use, including multi-vitamin/ mineral, herbal, plant or botanical, fish oil, and oil supplements, and not willing to discontinue before starting the study.
* Vegetarian or vegan diet
* Self-reported malabsorption or gastrointestinal issues
* Fruit and vegetable intake exceeding daily recommendations of 5 servings
* Smoking (vaping, conventional nicotine-containing products or marijuana)
* Current enrollee in a clinical research study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Microvascular Function | 4 weeks
  Microvascular function as measured by peripheral arterial tonometry (ENDO PAT 2000)

SECONDARY OUTCOMES:
Cytokines | 4 weeks
  Th17 cytokine panel
short chain fatty acids | 4 weeks
  both plasma and fecal
Bile acids | 4 weeks
  plasma bile acids
zonulin | 4 weeks
  serum zonulin
soluble lipopolysaccharide binding protein | 4 weeks
  plasma
cd14 | 4 weeks
  plasma
GLP-1 | 4 weeks
  fasting plasma levels
plasma lipids | 4 weeks
  total-, LDL-, HDL-cholesterol, and triglycerides
IGF/IGFbp | 4 weeks
  insulin like growth factor (IGF) and its associated binding proteins (BP)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta R Holt, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Academic Surge; Ragle Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No